CLINICAL TRIAL: NCT00450086
Title: Double-blind, Double-dummy, Randomised, Placebo-controlled, Multi-centre Phase III Clinical Study on the Efficacy and Tolerability of Budesonide Capsules vs. Mesalazine Granules vs. Placebo for Patients With Collagenous Colitis.
Brief Title: Budesonide Capsules vs. Mesalazine Granules vs. Placebo in Collagenous Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUC-60/COC; 2006-004159-39
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Collagenous Colitis
MeSH Terms: conditions — Colitis, Collagenous | interventions — Budesonide; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental)
  Interventions: Drug: Budesonide
- B (Experimental)
  Interventions: Drug: Mesalazine
- C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — 9 mg per day
  Arms: A
Drug: Mesalazine — 3 g per day
  Arms: B
Drug: Placebo — 0 g per day
  Arms: C

SUMMARY:
The purpose of this study is to determine whether budesonide or mesalazine is more active in the treatment of collagenous colitis.

DETAILED DESCRIPTION:
This study will check the reproducibility of the results reported in trials with budesonide in patients with collagenous colitis. Efficacy of mesalazine was never tested in collagenous colitis by placebo-controlled trials. This trial will check the superiority of mesalazine over placebo using the common clinical symptom of collagenous colitis, which is chronic or recurrent non-bloody, watery diarrhea.

ELIGIBILITY:
Inclusion Criteria (main):

* > 4 watery/soft stools on at least 4 days in the week prior to baseline
* > 3 stools per day on average within the last 7 days prior to baseline
* Symptoms (chronic watery diarrhea) for at least 3 months before baseline
* Complete colonoscopy within the last 12 weeks before baseline
* Histologically confirmed diagnosis of collagenous colitis

Exclusion Criteria:

* Evidence of infectious diarrhea
* Celiac disease
* Endoscopic-histologic findings, which may have caused diarrhea
* History of partial colonic resection
* Diarrhea as a result of the presence of other symptomatic organic disease of the gastrointestinal tract
* Active colorectal cancer or a history of colorectal cancer
* Severe co-morbidity substantially reducing life expectancy
* Abnormal hepatic function or liver cirrhosis (ALT, AST or AP >= 2 x ULN)
* Abnormal renal function (Cystatin C > ULN)
* Active peptic ulcer disease, local intestinal infection
* Asthma, diabetes mellitus, infection, osteoporosis, glaucoma, cataract, or cardiovascular disease if careful medical monitoring is not ensured
* Hemorrhagic diathesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-03; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission (<= 3 stools per day) after 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Rate of clinical remission (<= 3 stools per day) after 2 weeks | 2 weeks
Time to remission
Impact on stool consistency (watery/soft/solid) | 8 weeks
Impact on abdominal pain | 8 weeks
Impact on patient's general well-being | 8 weeks
Effect on histopathology | 8 weeks
Severity of diarrhea | 8 weeks
QoL | 8 weeks
PGA | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Miehlke, Professor, Principal Investigator — Center for digestive diseases
Locations (1):
- Center of digestive diseases, Hamburg, Germany

REFERENCES:
- [Result] Miehlke S, Madisch A, Kupcinskas L, Petrauskas D, Bohm G, Marks HJ, Neumeyer M, Nathan T, Fernandez-Banares F, Greinwald R, Mohrbacher R, Vieth M, Bonderup OK; BUC-60/COC Study Group. Budesonide is more effective than mesalamine or placebo in short-term treatment of collagenous colitis. Gastroenterology. 2014 May;146(5):1222-30.e1-2. doi: 10.1053/j.gastro.2014.01.019. Epub 2014 Jan 15. PMID 24440672